CLINICAL TRIAL: NCT01571102
Title: Study of Impact of Physiotherapy on Short-term Outcome After Meniscectomy.
Brief Title: Impact of Physiotherapy on Short-term Outcome After Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/161
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2014-12

CONDITIONS: Meniscectomy
MeSH Terms: interventions — Therapeutics; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- physiotherapy (Active Comparator): Promote mobility, strength and stability and exercises to reduce pain and swelling depending on the phase of tissue repair and evolution of the patient.
  Interventions: Behavioral: Therapy
- Rest (No Intervention)
- Home exercises (Active Comparator): Promote mobility, strength and stability and exercises to reduce pain and swelling depending on the phase of tissue repair and evolution of the patient.
  Interventions: Behavioral: Exercise therapy

INTERVENTIONS:
Behavioral: Therapy — week 1 - 4: 3 times/week, week 5 - 8: 2 times/week, duration 40min.
  Arms: physiotherapy
Behavioral: Exercise therapy — week 1 - 4: 3 times/week, week 5 - 8: 2 times/week, duration 30 min.
  Arms: Home exercises

SUMMARY:
In this study we investigate whether physiotherapy offers added value in rehabilitation after meniscectomy compared with no therapy or a home program. The population consists of 180 post-operative meniscus injury patients, operated at UZ Gent, the first 60 patients received no therapy, the next 60 patients were offered a treatment by their home physiotherapist according to our established protocol and the last 60 patients we have prepared a home program .

The physiotherapeutic treatment has been prepared based on scientific literature and own experience from the program at Ghent University and internships. It includes exercises to promote mobility, strength and stability and exercises to reduce pain and swelling depending on the phase of tissue repair and evolution of the patient. This schedule will be given to the patient along with the questionnaires at registration of the operation and will serve as a guideline for the physiotherapist for the rehabilitation of the patient after surgery. Monitoring of the evolution will take place by calling the physiotherapist on regular basis.

The home program is prepared on the basis of commonly used home exercises after arthroscopy and also includes exercises to promote mobility, strength and stability and exercises to reduce pain and swelling. The difference with the physiotherapeutic treatment is that there is no control and supervision of a physiotherapist and that the treatment is more limited. This program is given with the patient along with the questionnaires at registration of the operation.

Pre-operatively and 4 weeks, 3 months, 6 months and 12 months post-operatively, an evaluation of the current condition of the patient will happen on the basis of standardized questionnaires. Based on the results of these questionnaires, collected at different times, we can determine which treatment provides the best rehabilitation after meniscectomy. The first (preoperative) questionnaire, given at registration of the operation, is completed and given to the nurse of the day hospital on the day of surgery, the other (postoperative) questionnaires are sent electronically to the patient's email address and need to be returned, after filling up.

This study spends specific attention to the speed of resumption of work / sports and daily activities and the presence or absence of complaints.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative meniscectomy and surgery at Ghent University Hospital

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Speed of resumption of work/ sports and daily activities. | After 4 weeks post-operative
  This outcome will be derived from the VAS (Visual analogue scales) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 4 weeks post-operative
  This outcome will be derived from the KOOS (Knee injury and Osteoarthritis Outcome Score)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 4 weeks post-operative
  This outcome will be derived from the SF-36 (Short Form Health Survey 36) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 4 weeks post-operative
  This outcome will be derived from the Tegner questionnaire.
Speed of resumption of work/ sports and daily activities. | After 4 weeks post-operative
  This outcome will be derived from the FORSS (Factor Occupational Rating System Scale)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 4 weeks post-operative
  This outcome will be derived from a physiotherapeutic questionnaire.
Speed of resumption of work/ sports and daily activities. | After 3 months post-operative
  This outcome will be derived from the VAS (Visual analogue scales) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 3 months post-operative
  This outcome will be derived from the KOOS (Knee injury and Osteoarthritis Outcome Score)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 3 months post-operative
  This outcome will be derived from the SF-36 (Short Form Health Survey 36) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 3 months post-operative
  This outcome will be derived from the Tegner questionnaire.
Speed of resumption of work/ sports and daily activities. | After 3 months post-operative
  This outcome will be derived from the FORSS (Factor Occupational Rating System Scale)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 3 months post-operative
  This outcome will be derived from a physiotherapeutic questionnaire.
Speed of resumption of work/ sports and daily activities. | After 6 months post-operative
  This outcome will be derived from the VAS (Visual analogue scales) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 6 months post-operative
  This outcome will be derived from the KOOS (Knee injury and Osteoarthritis Outcome Score)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 6 months post-operative
  This outcome will be derived from the SF-36 (Short Form Health Survey 36) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 6 months post-operative
  This outcome will be derived from the Tegner questionnaire.
Speed of resumption of work/ sports and daily activities. | After 6 months post-operative
  This outcome will be derived from the FORSS (Factor Occupational Rating System Scale)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 6 months post-operative
  This outcome will be derived from a physiotherapeutic questionnaire.
Speed of resumption of work/ sports and daily activities. | After 1 year post-operative
  This outcome will be derived from the VAS (Visual analogue scales) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 1 year post-operative
  This outcome will be derived from the KOOS (Knee injury and Osteoarthritis Outcome Score)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 1 year post-operative
  This outcome will be derived from the SF-36 (Short Form Health Survey 36) questionnaire.
Speed of resumption of work/ sports and daily activities. | After 1 year post-operative
  This outcome will be derived from the Tegner questionnaire.
Speed of resumption of work/ sports and daily activities. | After 1 year post-operative
  This outcome will be derived from the FORSS (Factor Occupational Rating System Scale)questionnaire.
Speed of resumption of work/ sports and daily activities. | After 1 year post-operative
  This outcome will be derived from a physiotherapeutic questionnaire.
Speed of resumption of work/ sports and daily activities. | Pre-operative
  This outcome will be derived from the VAS (Visual analogue scales) questionnaire.
Speed of resumption of work/ sports and daily activities. | Pre-operative
  This outcome will be derived from the KOOS (Knee injury and Osteoarthritis Outcome Score)questionnaire.
Speed of resumption of work/ sports and daily activities. | Pre-operative
  This outcome will be derived from the SF-36 (Short Form Health Survey 36) questionnaire.
Speed of resumption of work/ sports and daily activities. | Pre-operative
  This outcome will be derived from the Tegner questionnaire.
Speed of resumption of work/ sports and daily activities. | Pre-operative
  This outcome will be derived from the FORSS (Factor Occupational Rating System Scale)questionnaire.
Speed of resumption of work/ sports and daily activities. | Pre-operative
  This outcome will be derived from a physiotherapeutic questionnaire.

SECONDARY OUTCOMES:
The presence of a total number of complaints. | pre-operative and 4 weeks, 3 months, 6 months and 1 year post-operative.
  This outcome will be derived from questionnaires: VAS, KOOS, SF-36, TEGNER, FORSS, physiotherapeutic questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be